CLINICAL TRIAL: NCT00018629
Title: Rehabilitation of Older Patients With Schizophrenia
Brief Title: Cognitive - Behavioral Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Granholm, Eric - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MHBS-043-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2008-09

CONDITIONS: Schizoaffective Disorder; Schizophrenia
Keywords: Aging; Neuropsychology; Psychotherapy; Rehabilitation; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

INTERVENTIONS:
Other:

SUMMARY:
The purpose of this study is to determine if Cognitive - Behavioral Social Skills Training (CBSST) improves functioning in older patients with schizophrenia.

DETAILED DESCRIPTION:
This is a randomized-control clinical trial. After completion the baseline assessment, subjects will be randomly assigned to either standard pharmacotherapy or SP+CBSST and will be followed for 18 months. The subjects will be 180 outpatients over the age of 45 with a diagnosis of schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

Patients must be 45 years of age or older with a diagnosis of schizophrenia or schizoaffective disorder.

Exclusion Criteria:

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2000-05; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Granholm, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States